CLINICAL TRIAL: NCT05212883
Title: Rapid Acceleration for Diagnostics in Underserved Populations: Home Testing
Brief Title: You and Me COVID Free
Acronym: YMCF
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00108149_1; 3U24MD016258-02S1 (NIH)
Record Dates: First submitted 2022-01-25; First posted 2022-01-28 (Actual); Results first posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: Rapid test; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Behavioral questionaires — Behavioral surveys and questionnaires

SUMMARY:
Observational, study that distributes rapid at-home, self-administered, SARS-CoV-2 antigen testing kits to households within pre-selected communities.

DETAILED DESCRIPTION:
This observational, cohort sub-study is embedded within a larger public health intervention that distributes at-home, self-administered, SARS-CoV-2 antigen testing kits to households within pre-selected communities through the CCPH. Within this sub-study, the investigators will evaluate the socio-behavioral mechanisms of SARS-CoV-2 community transmission, including social interactions, health behaviors, healthcare utilization, knowledge, disease burden, and feasibility of at-home testing. The central hypothesis is that focused community intervention will reduce COVID-19 transmission. The secondary hypothesis is that this intervention will increase vaccine uptake. Surveys and questionnaires will be completed by participants via a QR code from the test kits that directs participants to a link. Questionnaires will collect data on demographic characteristics, medical history and health status, COVID testing and symptoms, social interactions, knowledge of prevention strategies, infection risk, and attitudes towards vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Self- reported primary residence within the pre-identified communities
* Age >12 years at enrollment
* Provision of signed and dated informed consent form

Exclusion Criteria:

-None if above are met

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children >12 years of age living within pre-identified communities participating in the public health intervention
Sampling Method: Non-Probability Sample
Enrollment: 2778 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hornik, MD, PhD, MPH, Principal Investigator — Duke University
Locations (1):
- Merced County, Merced, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The project team utilized a robust communications campaign and mobilized community partners to assist with outreach and to organize COVID-19 (SARs-CoV-2) antigen testing kit distribution events. Community members received tests via in person at local distribution centers and events.
Groups:
- Behavioral Questionnaires: Questionnaires will collect data on demographic characteristics, medical history and health status, COVID testing and symptoms, social interactions, knowledge of prevention strategies, infection risk, and attitudes towards vaccines.
Period: Overall Study
Arm/Group | Behavioral Questionnaires
Started | 2778
Completed | 2653
Not Completed | 125
Not completed — Invalid test result | 125

BASELINE CHARACTERISTICS:
Population: Participants who completed the baseline questionnaire.
Arm/Group | Behavioral Questionnaires
Number analyzed (Participants) | 1001
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [29 to 50]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 687
  Male | 280
  Unknown or Not Reported | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 529
  Not Hispanic or Latino | 434
  Unknown or Not Reported | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 35
  Asian | 74
  Native Hawaiian or Other Pacific Islander | 5
  Black or African American | 39
  White | 546
  More than one race | 36
  Unknown or Not Reported | 266
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1001

OUTCOME MEASURES:

1. Primary Outcome: Main Reason for Testing for COVID-19
Description: Those that used a test from a kit were asked to provide the reason why they were doing a test. The possible answers are: "I wanted to be sure I/my child did not have COVID-19 before being around others", "I/my child had COVID-19 like symptoms", "I/my child was in close contact with someone who might have COVID-19", "I/my child was in close contact with someone who tested positive for COVID-19", "Someone in my household might have COVID-19", "Someone in my household tested positive for COVID-19", "Other"
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Questionnaires
Number analyzed (Participants) | 2778
Participants
  I wanted to be sure I/my child did not have COVID-19 before being around others | 1632
  I/my child had COVID-19 like symptoms | 493
  I/my child was in close contact with someone who might have COVID-19 | 238
  I/my child was in close contact with someone who tested positive for COVID-19 | 343
  Someone in my household might have COVID-19 | 118
  Someone in my household tested positive for COVID-19 | 152
  Other | 209
Statistical Analysis 1: Comparison: Behavioral Questionnaires; Comparison of the likelihood to test before gathering for age < 18 vs. age >= 18; Test type: Other; Odds Ratio (OR) = 1, 95% CI 2-sided [0.8 to 1.3]

2. Primary Outcome: Number of Positive COVID-19 Test Results
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Questionnaires
Number analyzed (Participants) | 2778
Participants | 269

3. Primary Outcome: Number of Participants Who Responded That They Have Received a COVID Vaccine
Time Frame: Baseline
Population: Participants who completed the baseline survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Questionnaires
Number analyzed (Participants) | 1001
Participants | 850

4. Secondary Outcome: Number of Participants Who Indicated That They Have Access to Necessary Personal Protective Equipment in Work Place
Time Frame: Baseline
Population: Participants who completed the baseline survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Questionnaires
Number analyzed (Participants) | 1001
Participants | 475

5. Secondary Outcome: Number of Participants Who Indicated They Have Tested Positive for COVID in Their Lifetime
Time Frame: Baseline
Population: Participants who completed the baseline survey and indicated having tested for COVID.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Questionnaires
Number analyzed (Participants) | 821
Participants | 237

6. Secondary Outcome: Number of Participants Who Report Knowing Where to Get COVID-19 Tests in the Community
Time Frame: Baseline
Population: Participants who completed the baseline survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Questionnaires
Number analyzed (Participants) | 1001
Participants | 757

7. Secondary Outcome: Number of Participants Who Report COVID Symptoms During Previous Week
Time Frame: Baseline
Population: Participants who completed the baseline survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Questionnaires
Number analyzed (Participants) | 1001
Participants | 627

8. Secondary Outcome: Likelihood of Future COVID-19 Vaccination
Description: Number of participants with front door survey entries indicating various levels of the likelihood the responder will get vaccinated in the future. Available options: "Very likely", "Somewhat likely", "Not very likely", "Not at all likely", and "Prefer not to answer".
Time Frame: Baseline
Population: Participants with front door survey entries that indicated the responder had not received a COVID-19 vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Questionnaires
Number analyzed (Participants) | 489
Participants
  Very likely | 119
  Somewhat likely | 140
  Not very likely | 59
  Not at all likely | 92
  Prefer not to answer/missing | 79

9. Secondary Outcome: Reasons for Not Getting a COVID-19 Vaccine
Description: Number of participants indicating various reasons for why they have not received a COVID-19 vaccine on the baseline survey. Available options: "I'm allergic to vaccines", "I don't like needles", "I'm not concerned about getting really sick from COVID-19", "I'm concerned about side effects from the vaccines", "I don't think vaccines work very well", "I don't trust that the vaccines will be safe", "I don't believe the COVID-19 pandemic is as bad as some people say it is", "I don't want to pay for it", and "I don't know enough about how well a COVID-19 vaccine works".
Time Frame: Baseline
Population: Participants who indicated they have not received a COVID-19 vaccine on the baseline survey. More than one answer can be selected by an individual participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Questionnaires
Number analyzed (Participants) | 121
Participants
  I'm allergic to vaccines | 5
  I don't like needles | 22
  I'm not concerned about getting really sick from COVID-19 | 3
  I'm concerned about side effects from the vaccines | 47
  I don't think vaccines work very well | 7
  I don't trust that the vaccines will be safe | 34
  I don't believe the COVID-19 pandemic is as bad as some people say it is | 4
  I don't want to pay for it | 3
  I don't know enough about how well a COVID-19 vaccine works | 16
  Other | 15

10. Secondary Outcome: Reasons for Getting a COVID-19 Vaccine
Description: Number of participants indicating various reasons for why they have received a COVID-19 vaccine on the baseline survey. Available options: "I want to keep my family safe", "I want to keep my community safe", "I want to keep myself safe", "I have a chronic health problem, like asthma or diabetes", "My doctor told me to get a COVID-19 vaccine", "I don't want to get really sick from COVID-19", "I want to feel safe around other people", "I believe life won't go back to normal until most people get a COVID-19 vaccine", "Required by my school or workplace", and "Required for travel".
Time Frame: Baseline
Population: Participants who indicated they have received a COVID-19 vaccine on the baseline survey. More than one answer can be selected by an individual participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Questionnaires
Number analyzed (Participants) | 850
Participants
  I want to keep my family safe | 712
  I want to keep my community safe | 477
  I want to keep myself safe | 557
  I have a chronic health problem, like asthma or diabetes | 135
  My doctor told me to get a COVID-19 vaccine | 86
  I don't want to get really sick from COVID-19 | 378
  I want to feel safe around other people | 404
  I believe life won't go back to normal until most people get a COVID-19 vaccine | 313
  Required by my school or workplace | 169
  Required for travel | 126
  Other | 24

11. Secondary Outcome: Perspective on Easiest Way to Obtain Free Oral COVID-19 Medications
Description: Number of front door survey entries indicating various ways in which participants would find it easy to get free COVID-19 oral medications. Available options: "An urgent care center". "A doctor's or other health professional's office", "A mobile health unit", "A drug store / pharmacy", "A grocery store", "A community center", "A place of worship", "A community park", "A neighborhood school", or "other". More than one answer can be selected by an individual participant.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Questionnaires
Number analyzed (Participants) | 2778
Participants
  An urgent care center | 503
  A doctor's or other health professional's office | 526
  A mobile health unit | 189
  A drug store / pharmacy | 1225
  A grocery store | 209
  A community center | 87
  A place of worship | 38
  A community park | 50
  A neighborhood school | 116
  Other | 25

12. Secondary Outcome: Method Used to Test for COVID-19
Description: Number of participants indicating the method used to test for COVID-19 on the baseline survey. Available options: "Nasal swab", "Throat swab", "Blood sample", and "Saliva".
Time Frame: Baseline
Population: Participants who indicated that they have tested for COVID-19.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Questionnaires
Number analyzed (Participants) | 821
Participants
  Nasal swab | 783
  Throat swab | 15
  Blood sample | 4
  Saliva | 17
  Missing | 2

ADVERSE EVENTS:
Time Frame: Adverse Event data was not collected.
Description: Adverse Event data was not collected.
Arm/Group | Behavioral Questionnaires
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-12-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT05212883/Prot_001.pdf
  • Statistical Analysis Plan (2022-04-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT05212883/SAP_002.pdf
  • Informed Consent Form (2021-12-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT05212883/ICF_000.pdf